CLINICAL TRIAL: NCT00435578
Title: An Open-Label, Phase 2 Study to Evaluate the Safety and Efficacy of Glufosfamide in the Treatment of Patients With Recurrent Sensitive Small Cell Lung Carcinoma
Brief Title: Safety and Efficacy Study of Glufosfamide in Patients With Recurrent Sensitive Small Cell Lung Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Threshold Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-304
Record Dates: First submitted 2007-02-13; First posted 2007-02-15 (Estimated); Last update posted 2009-04-30 (Estimated); Status verified 2009-04

CONDITIONS: Carcinoma, Small Cell Lung
Keywords: Recurrent Sensitive Small-Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — beta-D-glucosylisophosphoramide mustard

INTERVENTIONS:
Drug: Glufosfamide

SUMMARY:
The primary objectives of this study are:

1. To evaluate the efficacy of glufosfamide in subjects with extensive recurrent sensitive small cell lung cancer (SCLC) as measured by objective response rate
2. To evaluate the safety of glufosfamide in subjects with extensive recurrent sensitive SCLC

The secondary objectives are:

1. To evaluate the efficacy of glufosfamide in subjects with extensive recurrent sensitive SCLC as measured by duration of response, progression-free survival and overall survival
2. To evaluate the pharmacokinetics of glufosfamide and isophosphoramide mustard (IPM)

The exploratory objectives of this trial are:

1. To evaluate the effect of glufosfamide on lung cancer symptoms
2. To evaluate the role of tumor cell glucose transporter expression on the efficacy of glufosfamide

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/IEC
* Documented extensive SCLC with progression occurring at least 60 days after completion of first-line therapy (sensitive disease)
* Measurable disease by RECIST criteria (at least one target lesion; no target lesion may have received radiotherapy within 6 weeks of study start)
* A minimum of 21 days between prior radiation therapy, immunotherapy, or other anti-tumor therapy and study entry
* Recovered from reversible toxicities of prior therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2
* Hemoglobin ≥ 9.0 g/dL, ANC ≥ 1,500/µL, platelets ≥ 100,000/µL
* Total bilirubin ≤ 1.5-fold ULN
* AST/ALT ≤ 2.5-fold ULN (≤ 5-fold ULN if liver metastases)
* Creatinine clearance ≥ 60 mL/min (calculated by Cockcroft-Gault formula)
* All women of childbearing potential and all men must agree to use effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) from entry into the study through 6 months after the last dose

Exclusion Criteria:

* More than one previous chemotherapy regimen
* Concomitant or planned hormonal therapy, radiation therapy, biologic therapy, chemotherapy or other systemic antitumor therapy for SCLC other than protocol therapy
* Limited stage SCLC (defined as confined to one hemithorax including ipsilateral supraclavicular lymph nodes and excluding pleural effusion)
* Symptomatic brain metastases requiring corticosteroids
* Active clinically significant infection requiring antibiotics
* Known HIV positive or active hepatitis B or C
* Recent (one year) history or symptoms of cardiovascular disease (NYHA Class 2, 3, or 4), particularly coronary artery disease, arrhythmias or conduction defects with risk of cardiovascular instability, uncontrolled hypertension, clinically significant pericardial effusion, congestive heart failure, or stroke
* Other active malignancies (other than treated non-melanoma skin cancer or treated in situ cancer) within the past 5 years
* Major surgery within 28 days of the start of study treatment, without complete recovery
* Females who are pregnant or breast-feeding
* Participation in an investigational drug or device study within 28 days of the first day of dosing on this study
* Concomitant disease or condition that could interfere with the conduct of the study, or that, in the opinion of the investigator, could pose an unacceptable risk to the subject in this study.
* Unwillingness or inability to comply with the study protocol for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Bepler, MD, PhD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; John C Ruckdeschel, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute; Peter D Eisenberg, MD, Principal Investigator — California Cancer Center
Locations (3):
- United States (3):
  - California Cancer Center, Greenbrae, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Karmanos Cancer Institute, Detroit, Michigan